CLINICAL TRIAL: NCT07200531
Title: Impact of Biopsychosocial Psychotherapy Intervention on Maternal Life-Course Trauma and the Gut Microbiome
Brief Title: Does Psychotherapy Change the Gut Microbiome in Women of Child-bearing Age?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Responsible Party: Principal Investigator, Tiffany Moore, Associate Professor, University of Nebraska
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0613-25-EP
Record Dates: First submitted 2025-08-23; First posted 2025-10-01 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Chronic Stress
Keywords: Gut Microbiome; Life-course trauma; Psychotherapy
MeSH Terms: interventions — Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Psychotherapy Intervention (Experimental)
  Interventions: Behavioral: Psychotherapy

INTERVENTIONS:
Behavioral: Psychotherapy — 6-week psychotherapy group intervention

SUMMARY:
The goal of this clinical trial is to learn if group therapy for six weeks changes the gut microbiome in women. The main questions it aims to answer are:

Is chronic stress associated with the gut microbiome? Will six weeks of therapy change the gut microbiota?

Participants will:

Answer questionnaires about chronic stress Mail a stool sample before and after the intervention. Participate in a 1-hour group therapy session over the course of six weeks.

ELIGIBILITY:
Inclusion Criteria:

* Women over the age of 19 and less than 54. Able to understand/read English

Exclusion Criteria:

* Pregnant women and breast-feeding women Women who are actively participating in psychotherapy on a regular basis

Ages: 19 Years to 54 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Depression, Anxiety, and Stress Scales | 6 weeks
  Self-report mood disorder questionnaire
Perceived Stress | 6 weeks
  self-report questionnaire of perceived stress

CONTACTS AND LOCATIONS:
Overall Officials: Ashley J Blount, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No
This is a small pilot study.